CLINICAL TRIAL: NCT03787485
Title: Linking Individual Needs to Community and Clinical Services
Acronym: LINKS
Status: Completed | Type: Observational
Sponsor: Abby Lohr (Other)
Collaborators: Pima County Health Department (Unknown); Yuma County Health District (Unknown); El Rio Community Health Center (Other); Sunset Community Health Center (Unknown); Mariposa Community Health Center (Unknown); Arizona Community Health Outreach Workers Association (AzCHOW) (Unknown)
Responsible Party: Sponsor-Investigator, Abby Lohr, Senior Research Specialist, University of Arizona
Organization: University of Arizona (Other)
Other Study IDs: 1612044741R001
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Chronic Disease
Keywords: Community Health Worker; Community Clinical Linkage
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LINKS Participants: Study participants who took part in the LINKS intervention.
  Interventions: Behavioral: LINKS
- Electronic Medical Record Controls: The principal analytical strategy is propensity score matching, which will lead to the generation of a natural control group from the health centers existing electronic medical records. Propensity matching is highly effective in addressing selection bias of known confounders and enables causal inferences when randomization is not possible, feasible or appropriate, by creating matched groups with similar covariate distributions. Matched controls will be extracted from the electronic medical record from the participating clinics.

INTERVENTIONS:
Behavioral: LINKS — The primary aim of LINKS is to create community-clinical linkages between three community health centers and their respective county health departments in southern Arizona. This study will also develop and evaluate a chronic disease and emotional well-being intervention that will connect clinic patients to community-centered, county-delivered, community health worker programs.
  Groups: LINKS Participants

SUMMARY:
For 15 years, the Centers for Disease Control and Prevention (CDC)-funded Arizona Prevention Research Center (AzPRC) has been engaged in academic community collaborative research to reduce chronic disease health disparities among the Latino border communities in Arizona, which positions the center well to contribute to CDC's current winnable battle of nutrition, physical activity and obesity. The AzPRC's research study Linking Individual Needs to Community and Clinical Services (LINKS) will implement and evaluate a CHW-delivered preventive program linking primary care settings dedicated to reaching the under-served with community services that are county-delivered or -based. By developing community-clinical linkages, the AzPRC will help ensure access to, and quality of, culturally relevant prevention and promotion efforts. These efforts will result in a sustainable and scalable CHW model program that reduces obesity and associated chronic disease, and improves overall health in under-served communities at the Arizona U.S.-Mexico border.

DETAILED DESCRIPTION:
Over the past 15 years, CDC-funded AzPRC researchers have strengthened collaborations with community partners while developing and implementing comprehensive diabetes prevention and control programs (1998-2019), and policy intervention research (2009-2014) in Southern Arizona border communities. The community health worker (CHW)-led diabetes programs were successful in terms of community perception and health improvements. Despite this success, disparities in chronic disease remained unacceptably high. The investigators developed and implemented an innovative intervention research project, Acción Para La Salud (Acción), which engaged CHWs in community-level advocacy to empower border communities to address root causes of chronic disease. This community-based participatory research (CBPR) project recognized the importance of addressing the social determinants of health to overcome health disparities in chronic disease. The investigators have published results and processes of Acción.

Chronic disease and obesity health disparities continue to disproportionately affect Hispanic populations along the U.S. Mexico border in part due to barriers to healthful nutrition, adequate physical activity, and mental/emotional well-being as well as insufficient access to culturally appropriate health care services. In collaboration with our border-wide Community Action Board (CAB), the investigators are taking our intervention expertise one step further by developing and testing novel CHW-led interventions that will link community and clinical services.

In recent years, federally qualified community health centers (FQHCs), a major backbone of the primary care system in reaching under-served populations across the US, have begun to involve the CHW model into various services, often with a focus on chronic disease prevention and control. While CHWs help improve the quality and cultural relevancy of health care, improve patient centered care, and improve linkages between primary care and community services, each clinic adapts practices within their clinic environment without clear guidelines about best practices, or concrete evidence regarding activities best shown to lead to improvement in health outcomes. In addition, there may not be clear linkages from the clinic to CHW programs in the community that have been shown to be effective in chronic disease control and prevention, and there are challenges in identifying mechanisms for the sustainability of effective clinical or community programs. Our intervention research proposes to fill these gaps by establishing clear guidance and best practices for CHW involvement in primary care and community settings to prevent and manage chronic disease, and to promote mental/emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have pre-diabetes, glucose intolerance or diabetes, and/or hypertension, and/or high cholesterol
* Participants not receiving palliative care;
* Participants without a history of serious mental illness (SMI)
* Participants who are not pregnant;
* Participants who speak either English or Spanish;
* Participants who are geographically close to the community based site; and
* Participants who consent to participate in the study.

Exclusion Criteria:

* Participants who do not consent to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be adults (21 and older), among whom approximately 70% are expected to be women, and the majority (at least 60%) to be Hispanic.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change from past (three years to baseline) participant glycosylated hemoglobin on the A1c test reported in electronic medical record after initiation of intervention | July 14, 2014- June 30, 2019
  Glycosylated hemoglobin (mmol/mol) will be extracted from laboratory reports reported in the electronic medical record.
Change from past (three years to baseline) participant body mass index (BMI) calculated from height (meters) and weight in (kilograms) reported in electronic medical record after initiation of intervention | July 14, 2014- June 30, 2019
  Height and weight reported in the participant's electronic medical record will be combined to report BMI in kg/m^2.
Change from past (three years to baseline) participant blood pressure based on systolic and diastolic blood pressures reported in electronic medical record after initiation of intervention | July 14, 2014- June 30, 2019
  Systolic and diastolic blood pressure (mmHg) will be extracted from vitals reported in the participant's electronic medical record.
Change from past (three years to baseline) participant total cholesterol as measured by low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglycerides reported in electronic medical record after initiation of intervention | July 14, 2014- June 30, 2019
  LDL, HDL, and triglycerides (mg/dL) reported in the participant's electronic medical record will be combined to report total cholesterol (mg/dL).

SECONDARY OUTCOMES:
Change from baseline in participant self-rated health, emotional well-being, and life satisfaction on 3 questions from the Behavioral Risk Factor Surveillance System (BRFSS) at 3 and 6 months | July 14, 2017-March 30, 2019
  The investigators will ask three questions from the BRFSS:
  1. Would you say in general your health is: (Excellent / Very good / Good / Fair / Poor)
  2. How often do you get the social and emotional support you need? (Always / Usually / Sometimes / Rarely / Never)
  3. In general, how satisfied are you with your life? (Very satisfied / Satisfied / Dissatisfied / Very Dissatisfied)
  Responses from the BRFSS are Likert type questions. Individual items from the scales will be tabulated and summarized at each administration of the questionnaire. The outcome at each timepoint for a given subject on a given scale will be the sum of the scores of the items from that scale. An increase in the score demonstrates a positive outcome.
Change from baseline in participant physical activity frequency in the last week on 1 question physical activity question at 3 and 6 months | July 14, 2017-March 30, 2019
  To determine participant physical activity, the investigators will ask a single question regarding the amount of physical activity the subject engaged in during the previous week:
  In the past week, on how many days have you done a total of 30 minutes or more of physical activity, which was enough to raise your breathing rate? (0-7 days)
  An increase in days reported demonstrates a positive outcome.
Change from baseline in participant mental and physical health on Short Form 8 Health Assessment (SF8) at 3 and 6 months | July 14, 2017-September 30, 2019
  Responses from the SF8 are Likert type questions. Individual items from this scale will be tabulated and summarized at each administration of the questionnaire. The outcome at each timepoint for a given subject on a given scale will be the sum of the scores of the items from that scale. An increase in the score demonstrates a positive outcome.
Change from baseline in participant social support on the Social Support Inventory (Enhancing Recovery in Coronary Heart Disease, ENRICHED) (SSI) at 3 and 6 months | July 14, 2017-September 30, 2019
  Responses from the SSI scales are Likert type questions, with the exception of SSI question 7 (Are you currently married or living with a partner? Yes/No). Individual items from this scale will be tabulated and summarized at each administration of the questionnaire. The outcome at each timepoint for a given subject on a given scale will be the sum of the scores of the items from that scale (excluding SSI question 7). An increase in the score demonstrates a positive outcome.
Change from baseline in participant hope on the State Hope Scale (SHS) at 3 and 6 months | July 14, 2017-September 30, 2019
  A total score for the SHS can be obtained by adding the values of the responses to each item, yielding a score from 6 - 48. An increase in the score demonstrates a positive outcome.
Change from baseline in participant depression on the Center for Epidemiologic Studies Depression Scale (CES-D-R 10) at 3 and 6 months | July 14, 2017-September 30, 2019
  A total score for the CES-D-R 10 scale is found by determining the sum of the items which are scored as:
  Rarely or none of the time (less than 1 day); Some or a little of the time (1 - 2 days); Occasionally or a moderate amount of time (3 - 4 days); All of the time (5 - 7 days)
  Questions 5 & 8: Rarely or none of the time (less than 1 day) = 3 to All of the time (5 - 7 days) = 0
  All other questions: Rarely or none of the time (less than 1 day) = 0 to All of the time (5 - 7 days) = 3
  An increase in the score demonstrates a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Carvajal, PhD, MPH, Principal Investigator — University of Arizona Prevention Research Center
Locations (5):
- United States (5):
  - Mariposa Community Health Center, Nogales, Arizona
  - El Rio Community Health Center, Tucson, Arizona
  - Pima County Health Department, Tucson, Arizona
  - Sunset Community Health Center, Yuma, Arizona
  - Yuma County Health District, Yuma, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohr AM, Ingram M, Nunez AV, Reinschmidt KM, Carvajal SC. Community-Clinical Linkages With Community Health Workers in the United States: A Scoping Review. Health Promot Pract. 2018 May;19(3):349-360. doi: 10.1177/1524839918754868. Epub 2018 Jan 24. PMID 29363334
- [Background] Ingram M, Doubleday K, Bell ML, Lohr A, Murrieta L, Velasco M, Blackburn J, Sabo S, Guernsey de Zapien J, Carvajal SC. Community Health Worker Impact on Chronic Disease Outcomes Within Primary Care Examined Using Electronic Health Records. Am J Public Health. 2017 Oct;107(10):1668-1674. doi: 10.2105/AJPH.2017.303934. Epub 2017 Aug 17. PMID 28817321
- [Background] Reinschmidt KM, Ingram M, Morales S, Sabo SJ, Blackburn J, Murrieta L, David C, Carvajal SC. Documenting Community Health Worker Roles in Primary Care: Contributions to Evidence-Based Integration Into Health Care Teams, 2015. J Ambul Care Manage. 2017 Oct/Dec;40(4):305-315. doi: 10.1097/JAC.0000000000000178. PMID 28350634
- [Derived] Lohr AM, Ingram M, Carvajal SC, Doubleday K, Aceves B, Espinoza C, Redondo F, Coronado G, David C, Bell ML. Protocol for LINKS (linking individual needs to community and clinical services): a prospective matched observational study of a community health worker community clinical linkage intervention on the U.S.-Mexico border. BMC Public Health. 2019 Apr 11;19(1):399. doi: 10.1186/s12889-019-6725-1. PMID 30975126